CLINICAL TRIAL: NCT05935683
Title: Rhinosinusitis Italian Network (RINET): the Italian Registry for Severe, Uncontrolled Chronic Rhinosinusitis
Brief Title: Rhinosinusitis Italian Network: the Italian Registry for Severe, Uncontrolled Chronic Rhinosinusitis
Acronym: RINET
Status: Recruiting | Type: Observational
Sponsor: Italian Academy of Rhinology (Other)
Collaborators: Accademia Italiana di Citologia Nasale (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2876
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis
Keywords: chronic rhinosinusitis with nasal polyps; chronic rhinosinusitis without nasal polyps; Otorhinolaryngologic Diseases; Respiratory Tract Diseases; Paranasal Sinus Diseases; Sinusitis; Nose Diseases; chronic rhinosinusitis (diagnosis)
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Respiratory Tract Diseases; Paranasal Sinus Diseases; Sinusitis; Nose Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Severe Uncontrolled Chronic Rhinosinusitis patients (CRS) — Obsertvation
  Other Names: Adult chronic rhinosinusitis patients.

SUMMARY:
This observatory aims to collect, as widely as possible, the Italian cases of patients with uncontrolled CRS. Patient will be enrolled by the centers of the Italian Network of Rhinosinusitis (Rhinosinusitis Italian Network: RINET), and they will be treated using a multidisciplinary team approach (allergists, otolaryngologists and pneumologists) in a real-world clinical set-up.

This real-life chronic rhinosinusitis registry aims at longitudinal data collection from patients attending specialist care centres across Italy.

DETAILED DESCRIPTION:
The primary objectives of the study are:

* to characterize and to describe the evolution of uncontrolled Chronic Rhinosinusitis (CRS);
* to facilitate and to characterize the phenotyping and endotyping of CRS;
* studying the efficacy and safety of the principal therapeutic strategies and approaches to uncontrolled CRS in real-life;
* supporting the development of diagnostic methodologies and innovative therapeutic strategies for CRS;
* to evaluate the clinical and economic-health impact of the different therapeutic approaches (including systemic corticosteroids) used for uncontrolled CRS;
* to describe factors associated with therapeutic choices and how much this factors influence natural history of the CRS;
* Studying and identifying biomarkers and predictors of response to different therapies;
* to increase the "awareness" of CRS in patients, in public opinion, in the national and international scientific community, and in the Italian clinical community of the otolaryngologists, the allergists and the pneumologists.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of bilateral Chronic Rhinosinusitis that have at least three (in case of patients previously treated with surgical approaches) or four (in case of patients never treated with nasal sinus surgery) of the following criteria:

  * Evidence of type 2 inflammation (at least 250 blood eosinophils per microliter and / or at least 10 eosinophils / HPF from a histological sample of sinus mucosa and / or at least one finding of moderate eosinophilia on nasal cytology and / or total serum IgE >100 IU / ml);
  * at least two Short courses of systemic corticosteroids or lorg-term Systemic Corticosteroids therapy for Chronic Rhinosinusitis;
  * Significant deterioration in the quality of life (Sinonasal Outcome Test 22 - SNOT-22>= 40 and / or Visual Analogue Scale - Global VAS of symptoms>= 5);
  * Loss of Smell (VAS for hyposmia> = 7)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Severe, Uncontrolled Chronic Rhinosinusitis with or without nasal polyps according to the European Position Paper on Rhinosinusitis and Nasal Polyps - EPOS2020 and to the EUFOREA consensus on biologics for CRSwNP with or without asthma
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2031-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score | Every year to ten year
  Change from baseline in total Nasal Polyp Score at year 1 to ten. The Nasal Polyp Score is the sum of the right and left nostril scores (maximum 8), as evaluated by nasal endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Marco Heffler, MD, PhD, Study Chair — Personalized Medicine, Asthma and Allergy - IRCCS Humanitas Research Hospital, Rozzano, Italy
Locations (1):
- Personalized Medicine, Asthma and Allergy - IRCCS Humanitas Research Hospital, Rozzano, MIlan, Italy

REFERENCES:
- [Background] Fokkens WJ, Lund V, Bachert C, Mullol J, Bjermer L, Bousquet J, Canonica GW, Deneyer L, Desrosiers M, Diamant Z, Han J, Heffler E, Hopkins C, Jankowski R, Joos G, Knill A, Lee J, Lee SE, Marien G, Pugin B, Senior B, Seys SF, Hellings PW. EUFOREA consensus on biologics for CRSwNP with or without asthma. Allergy. 2019 Dec;74(12):2312-2319. doi: 10.1111/all.13875. Epub 2019 Jul 15. PMID 31090937
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- See also: Description Rhinosinusitis Italian NETwork — http://rinet-registry.org/